CLINICAL TRIAL: NCT04635631
Title: AN OPEN-LABEL, SINGLE-ARM, PHASE 1 STUDY OF PHARMACOKINETICS, SAFETY AND ANTI-TUMOR ACTIVITY OF TALAZOPARIB MONOTHERAPY IN CHINESE PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: STUDY OF TALAZOPARIB MONOTHERAPY IN CHINESE PARTICIPANTS WITH ADVANCED SOLID TUMORS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3441049
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- talazoparib (Experimental): 1 mg QD
  Interventions: Drug: talazoparib

INTERVENTIONS:
Drug: talazoparib — Talazoparib will be administered orally on a continuous basis. Each cycle will consist of 28 days.

SUMMARY:
A phase1 study to evaluate the PK (single dose and multiple doses) and safety of talazoparib 1 mg Once Daily in Chinese adult participants with advanced solid tumors. A maximum of approximately 15 participants will be enrolled such that approximately 12 evaluable participants complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of locally advanced or metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available.
* ECOG Performance Status 0 or 1.
* Adequate Bone Marrow, Renal and Liver Function.

Exclusion Criteria:

* Participants with brain metastases.
* Current or anticipated use of P gp inhibitor and/or inducer within 7 days prior to study intervention from lead-in to end of Cycle 1; concomitant use of potent P gp inhibitor after Cycle 1 until the end of treatment.
* Prior treatment with a PARP inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Luo Y, Cheng Y, Wu C, Ye H, Chen N, Zhang F, Wei H, Xu B. Pharmacokinetics, safety, and antitumor activity of talazoparib monotherapy in Chinese patients with advanced solid tumors. Invest New Drugs. 2023 Jun;41(3):503-511. doi: 10.1007/s10637-023-01351-w. Epub 2023 May 12. PMID 37171721
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 15 participants were enrolled and received talazoparib 1 mg once daily (QD).
Groups:
- Talazoparib 1 mg QD: Participants received a single oral dose of talazoparib 1mg on Day -9 (lead-in dose), and then received talazoparib 1mg QD in 28-day cycles (maximum 9 cycles), starting from Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Talazoparib 1 mg QD
Started | 15
Completed | 0
Not Completed | 15
Not completed — Adverse Event | 1
Not completed — Progressive disease | 13
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants who received at least one dose of study intervention.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 53 [31 to 72]
Age, Customized [Count of Participants; unit: Participants]
  18 to <45 years | 4
  45 to <65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 15
  Other (Not Chinese) | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Talazoparib Following Single Oral Dose
Description: Maximum plasma concentration of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9. Cmax was directly observed from data.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 96 hours, 168 hours and 216 hours post Day -9 dosing
Population: The analysis population included all participants enrolled and treated who had at least 1 of the pharmacokinetic (PK) parameters of interest in the single-dose and/or multiple dose PK part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Talazoparib 1 mg Once Daily (QD): Participants received a single oral dose of talazoparib 1mg on Day -9 (lead-in dose), and then received talazoparib 1 mg QD in 28-day cycles (maximum 9 cycles), starting from Cycle 1 Day 1. Participants entered follow-up phase at least 28 days and no more than 35 days after last dose/discontinuation of study treatment.
Arm/Group | Talazoparib 1 mg Once Daily (QD)
Number analyzed (Participants) | 15
nanogram/milliliter (ng/mL) | 8.506 (41)

2. Primary Outcome: Time to Cmax (Tmax) of Talazoparib Following Single Oral Dose
Description: Time to reach Cmax (maximum plasma concentration) of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9.
Time Frame: as for outcome 1
Population: The analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of interest in the single-dose and/or multiple dose PK part.
Measure: Median (Full Range); unit: hours
Groups:
- Talazoparib 1mg QD: Participants received a single oral dose of talazoparib 1mg on Day -9 (lead-in dose), and then received talazoparib 1mg QD in 28-day cycles (maximum 9 cycles), starting from Cycle 1 Day 1. Participants entered follow-up phase at least 28 days and no more than 35 days after last dose/discontinuation of study treatment.
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
hours | 1.90 [0.517 to 7.63]

3. Primary Outcome: Area Under Plasma Concentration-Time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Talazoparib Following Single Oral Dose
Description: Area under the plasma concentration versus time curve from time zero to the time of the last quantifiable concentration of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
ng*hr/mL | 172.0 (32)

4. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time Tau (AUCtau) of Talazoparib Following Single Oral Dose
Description: Area under the plasma concentration versus time curve from time zero to the time tau (=24 hours) of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
ng*hr/mL | 86.54 (29)

5. Primary Outcome: Apparent Oral Clearance (CL/F) of Talazoparib Following Single Oral Dose
Description: Apparent oral clearance of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F is calculated as dose/AUCinf. AUCinf = area under the plasma concentration versus time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 1
Population: The analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in the single-dose and/or multiple dose PK part. Number of participants analyzed = number of participants in the analysis population that contributed to the summary statistics of this outcome measure (OM).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/hr)
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 10
liter/hour (L/hr) | 4.798 (31)

6. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Talazoparib Following Single Oral Dose
Description: Apparent volume of distribution of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9. Vz/F is calculated as Dose/(AUCinf * kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUCinf is area under the plasma concentration versus time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 1
Population: The analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in the single-dose and/or multiple dose PK part. Number of participants analyzed = number of participants in the analysis population that contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 10
Liter | 456.8 (37)

7. Primary Outcome: Terminal Half-Life (t1/2) of Talazoparib Following Single Oral Dose
Description: Terminal half-life of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9. t1/2 is defined as the time for plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 10
hours | 67.00 (11.779)

8. Primary Outcome: Area Under Plasma Concentration-Time Profile From Time Zero to Infinity (AUCinf) of Talazoparib Following Single Oral Dose
Description: Area under the plasma concentration versus time curve from time zero extrapolated to infinite time of talazoparib after the participant received a single oral lead-in dose of talazoparib 1 mg on Study Day -9.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 10
ng*hr/mL | 208.3 (31)

9. Primary Outcome: Cmax of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Maximum plasma concentration of talazoparib at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: The analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in the single-dose and/or multiple dose PK part. Number of participants analyzed = number of participants in the analysis population that contributed data to this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
ng/mL | 14.35 (169)

10. Primary Outcome: Tmax of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Time for Cmax of talazoparib at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
hours | 1.85 [0.533 to 23.7]

11. Primary Outcome: Minimum Plasma Concentration (Cmin) of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Minimum plasma concentration observed during the dosing interval at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
ng/mL | 2.616 (95)

12. Primary Outcome: AUCtau of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Area under the plasma concentration versus time curve within a dosing interval of tau (=24 hours) at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
ng*hr/mL | 147.8 (123)

13. Primary Outcome: CL/F of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Apparent clearance at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is a quantitative measure of the rate at which a drug substance is removed from the blood. Steady-state CL/F is calculated as dose/AUCtau. AUCtau = area under the plasma concentration versus time curve within a dosing interval of tau (=24 hours) at steady state after multiple doses.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
L/hr | 6.770 (123)

14. Primary Outcome: Observed Accumulation Ratio (Rac) of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Observed accumulation ratio at steady state after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22. Rac is calculated as AUCtau/AUCsd,tau, where AUCtau = Area under the plasma concentration versus time curve within a dosing interval of tau (=24 hours) at steady state after multiple doses, AUCsd,tau = area under the plasma concentration versus time curve from time zero extrapolated to the time tau (=24 hours) after single dose.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 12
ratio | 1.733 (127)

15. Primary Outcome: Steady-State Accumulation Ratio (Rss) of Talazoparib Following Multiple Oral Doses (Steady State)
Description: Steady-state accumulation ratio after the participant received multiple oral doses of talazoparib 1 mg QD from Cycle 1 Day 1 to Cycle 1 Day 22. Rss is calculated as AUCtau/AUCinf, where AUCtau = Area under the plasma concentration versus time curve within a dosing interval of tau (=24 hours) at steady state after multiple doses, AUCinf = Area under the plasma concentration versus time curve from time zero extrapolated to infinite time after single dose.
Time Frame: Pre-dose and 0.5 hours, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours after dosing on Cycle 1 Day 22.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 8
ratio | 0.6958 (192)

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs with start date during the on-treatment period (including on the date of first dose). Grades of AEs were defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03. Grade 1(mild)=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2(moderate)=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE. Treatment-related TEAEs were determined by the investigator.
Time Frame: Baseline (the latest non-missing value prior to or on the date of first dose of talazoparib) to at least 28 days after the last dose of talazoparib (maximum of approximately 46 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  All-causality TEAEs | 14
  Treatment-related TEAEs | 13
  Grade 3 or 4 all-causality TEAEs | 10
  Grade 3 or 4 treatment-related TEAEs | 6
  Grade 5 TEAEs (TEAEs leading to death) | 0
  All-causality TEAEs leading to dose interruption of talazoparib | 3
  Treatment-related TEAEs leading to dose interruption of talazoparib | 2
  All-causality TEAEs leading to dose reduction of talazoparib | 5
  Treatment-related TEAEs leading to dose reduction of talazoparib | 5
  All-causality TEAEs leading to discontinuation from talazoparib | 1
  Treatment-related TEAEs leading to discontinuation from talazoparib | 1

17. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect. Treatment-related SAEs were determined by the investigator.
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  All-causality SAE | 3
  Treatment-related SAE | 3

18. Secondary Outcome: Number of Participants With Grade 3 or 4 All-Causality TEAEs by Preferred Term (PT) and Maximum CTCAE Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs with start date during the on-treatment period (including on the date of first dose). Grades of AEs were defined by NCI CTCAE version 4.03. Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated. Treatment-related TEAEs were determined by the investigator. Grade 3 or 4 TEAEs reported by at least 1 participant are reported here.
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Grade 3 Gamma-glutamyltransferase increased | 3
  Grade 4 Gamma-glutamyltransferase increased | 1
  Grade 3 Anaemia | 4
  Grade 3 Neutrophil count decreased | 3
  Grade 4 Neutrophil count decreased | 1
  Grade 3 Platelet count decreased | 1
  Grade 4 Platelet count decreased | 2
  Grade 3 Aspartate aminotransferase increased | 2
  Grade 3 Abdominal distension | 1
  Grade 3 Blood bilirubin increased | 1
  Grade 3 Hypercholesterolaemia | 1
  Grade 3 Hyperglycaemia | 1
  Grade 4 Hypernatraemia | 1
  Grade 4 Hyperuricaemia | 1
  Grade 3 Hypokalaemia | 1
  Grade 3 Hyponatraemia | 1
  Grade 3 Neutropenia | 1

19. Secondary Outcome: Number of Participants With Grade 3 or 4 Treatment-Related TEAEs by PT and Maximum CTCAE Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs with start date during the on-treatment period (including on the date of first dose). Grades of AEs were defined by NCI CTCAE version 4.03. Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated. Treatment-related TEAEs were determined by the investigator. Grade 3 or 4 treatment-related TEAEs reported by at least 1 participant are reported here.
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Grade 3 Anaemia | 4
  Grade 3 Neutrophil count decreased | 3
  Grade 4 Neutrophil count decreased | 1
  Grade 3 Platelet count decreased | 1
  Grade 4 Platelet count decreased | 2
  Grade 3 Hyponatraemia | 1
  Grade 3 Neutropenia | 1

20. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Interruption of Talazoparib by PT
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=AEs with start date during the on-treatment period (including on the date of first dose). Treatment-related TEAEs were determined by the investigator.
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  All-causality Anaemia leading to dose interruption | 1
  Treatment-related Anaemia leading to dose interruption | 1
  All-causality Aspartate aminotransferase increased leading to dose interruption | 1
  All-causality Neutrophil count decreased leading to dose interruption | 1
  Treatment-related Neutrophil count decreased leading to dose interruption | 1
  All-causality Platelet count decreased leading to dose interruption | 1
  Treatment-related Platelet count decreased leading to dose interruption | 1

21. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Reduction of Talazoparib by PT
Description: as for outcome 20
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  All-causality Anaemia leading to dose reduction | 3
  Treatment-related Anaemia leading to dose reduction | 3
  All-causality Neutrophil count decreased leading to dose reduction | 3
  Treatment-related Neutrophil count decreased leading to dose reduction | 3
  All-causality Platelet count decreased leading to dose reduction | 3
  Treatment-related Platelet count decreased leading to dose reduction | 3
  All-causality Neutropenia leading to dose reduction | 1
  Treatment-related Neutropenia leading to dose reduction | 1
  All-causality Hypernatraemia leading to dose reduction | 1
  All-causality Hyponatraemia leading to dose reduction | 1
  Treatment-related Hyponatraemia leading to dose reduction | 1

22. Secondary Outcome: Number of Participants With TEAEs Leading to Discontinuation From Talazoparib by PT
Description: as for outcome 20
Time Frame: as for outcome 16
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  All-causality Neutrophil count decreased leading to discontinuation from talazoparib | 1
  Treatment-related Neutrophil count decreased leading to discontinuation from talazoparib | 1

23. Secondary Outcome: Number of Participants With On-Treatment Hematology Laboratory Abnormalities Shifting From <=Grade 2 at Baseline to Grade 3/4 Post-Baseline by Maximum CTCAE Grade
Description: Hematology lab parameters included hemoglobin, hematocrit, red blood cell (RBC) count, platelet count, white blood cell (WBC) count, neutrophils%, eosinophils%, monocytes%, basophils%, lymphocytes%. Grades of lab abnormalities were defined per NCI CTCAE version 4.03. Grade 1(mild)=asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2(moderate)=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL;Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; disabling limiting self-care ADL;Grade 4=life-threatening consequences, urgent intervention indicated. On-treatment is defined as time from first dose date of talazoparib through at least 28 days after last dose or start day of new anti-cancer therapy minus 1 day. Shifts meeting criteria and reported in at least 1 participant are reported in this OM.
Time Frame: From first dose date up to at least 28 days after last dose or to the start of new anti-cancer drug therapy minus 1 day (whichever was earlier) (maximum of approximately 46 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Anemia: Grade 0 to Grade 3 | 3
  Anemia: Grade 1 to Grade 3 | 1
  Lymphocyte count decreased: Grade 0 to Grade 3 | 1
  Neutrophil count decreased: Grade 0 to Grade 3 | 5
  Neutrophil count decreased: Grade 0 to Grade 4 | 1
  Platelet count decreased: Grade 0 to Grade 3 | 1
  Platelet count decreased: Grade 0 to Grade 4 | 2
  White blood cell decreased: Grade 0 to Grade 3 | 1

24. Secondary Outcome: Number of Participants With On-Treatment Chemistry Laboratory Abnormalities Shifting From <=Grade 2 at Baseline to Grade 3/4 Post-Baseline by Maximum CTCAE Grade
Description: Chemistry lab parameters included blood urea nitrogen or urea,creatinine,glucose (fasting),calcium,sodium,potassium,magnesium,chloride,aspartate aminotransferase,alanine aminotransferase,total bilirubin,alkaline phosphatase,uric acid,albumin,total protein,creatinine clearance. Grades of lab results were defined per NCI CTCAE v4.03.Grade 1=asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL;Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; disabling limiting self-care ADL;Grade 4=life-threatening consequences, urgent intervention indicated.On-treatment=time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day. Shifts meeting criteria and reported in at least 1 participant are reported.
Time Frame: as for outcome 23
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Alkaline phosphatase increased: Grade 0 to Grade 3 | 1
  Aspartate aminotransferase: Grade 1 to Grade 3 | 2
  Blood bilirubin increased: Grade 0 to Grade 3 | 1
  Hyperglycemia: Grade 1 to Grade 3 | 1
  Hypernatremia: Grade 0 to Grade 4 | 1
  Hypokalemia: Grade 0 to Grade 3 | 1
  Hyponatremia: Grade 0 to Grade 3 | 1

25. Secondary Outcome: Number of Participants With On-Treatment Urinalysis Laboratory Abnormalities Shifting From <=Grade 2 at Baseline to Grade 3/4 Post-Baseline by Maximum CTCAE Grade
Description: Urinalysis examined pH,glucose,protein,blood,ketones,nitrites,leukocyte esterase/leukocytes,urobilinogen,urine bilirubin,microscopy. Grades of lab results were defined by NCI CTCAE v4.03. Grade 1(mild)=asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2(moderate)=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL;Grade 3=severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; disabling limiting self-care ADL;Grade 4=life-threatening consequences, urgent intervention indicated. On-treatment=time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day. This OM is based only on lab data. Grade 4 proteinuria cannot be assessed based only on lab data, so is not applicable/not reported.
Time Frame: as for outcome 23
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention. Number of participants analyzed = number of participant evaluable for this OM.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 13
Participants
  Protenuria: Grade 0 to Grade 3 | 0
  Protenuria: Grade 1 to Grade 3 | 0
  Protenuria: Grade 2 to Grade 3 | 0

26. Secondary Outcome: Number of Participants With On-Treatment Vital Signs Data Meeting Pre-Specified Criteria for Potentially Clinically Significant Results
Description: Vital signs data included systolic and diastolic blood pressure (BP), pulse rate, respiratory rate (RR), temperature and weight. BP and pulse rate were recorded in sitting position. Potentially clinically significant vital signs abnormalities are defined as: systolic BP absolute result >180 mmHg and increase from baseline ≥40 mmHg, absolute result <90 mmHg and decrease from baseline >30 mmHg; diastolic BP absolute result >110 mmHg and increase from baseline ≥30 mmHg, absolute result <50 mmHg and decrease from baseline >20 mmHg, increase from baseline ≥20 mmHg; pulse rate absolute result >120 beats per minute (bpm) and increase from baseline >30 bpm, absolute result <50 bpm and decrease from baseline > 20 bpm; weight >10% decrease from baseline. Participants with vital signs data meeting any criteria above are reported in this OM if any. On-treatment is defined as time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day.
Time Frame: as for outcome 23
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants | 1

27. Secondary Outcome: Number of Participants With On-Treatment Maximum QT Interval (Bazett's Correction) (QTcB) and QT Interval (Fridericia's Correction) (QTcF) Data by Category
Description: Standard 12-lead electrocardiograms (ECGs) utilizing limb leads (with a 10 second rhythm strip) were collected using an ECG machine that automatically calculated the heart rate and measured PR, RR, QT intervals, QTc, QTcF and QRS complex. All scheduled ECGs were performed after the participant had rested quietly for at least 10 minutes. On-treatment is defined as the time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day.
Time Frame: as for outcome 23
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  QTcB interval value <=450 millisecond (msec) | 9
  QTcB interval value >450 msec and <=480 msec | 5
  QTcB interval value >480 msec and <=500 msec | 0
  QTcB interval value >500 msec | 1
  QTcF interval value <=450 msec | 14
  QTcF interval value >450 msec and <=480 msec | 1
  QTcF interval value >480 msec and <=500 msec | 0
  QTcF interval value>500 msec | 0

28. Secondary Outcome: Number of Participants With On-Treatment Maximum Increase From Baseline in QTcB and QTcF Data by Category
Description: as for outcome 27
Time Frame: as for outcome 23
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  QTcB interval increase from baseline <=30 msec | 9
  QTcB interval increase from baseline >30 msec and <=60 msec | 2
  QTcB interval increase from baseline >60 msec | 4
  QTcF interval increase from baseline <=30 msec | 9
  QTcF interval increase from baseline >30 msec and <=60 msec | 3
  QTcF interval increase from baseline >60 msec | 3

29. Secondary Outcome: Number of Participants With On-Treatment Concomitant Medications
Description: Concomitant medications or nondrug treatments/procedures were defined as medications or nondrug treatments/procedures, other than study intervention, which started prior to first dose date of study treatment and continued on on-treatment period as well as those started during the on-treatment period. On-treatment is defined as the time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day.
Time Frame: From first dose date up to at least 28 days after last dose/start day of new anti-cancer drug therapy minus 1 day (maximum of approximately 46 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants | 14

30. Secondary Outcome: Number of Participants With On-Treatment Concomitant Medications With Frequency >=20% by PT
Description: Concomitant medications or nondrug treatments/procedures were defined as medications or nondrug treatments/procedures, other than study intervention, which started prior to first dose date of study treatment and continued on on-treatment period as well as those started during the on-treatment period. On-treatment is defined as the time from first dose date through at least 28 days after last dose/start day of new anti-cancer therapy minus 1 day. On-treatment concomitant medications reported in at least 20% participants are reported for this OM.
Time Frame: as for outcome 29
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Recombinant human thrombopoietin | 3
  Lidocaine | 3
  Glucose | 3
  Dexamethasone sodium phosphate | 3
  Granulocyte colony stimulating factor | 3
  Herbal preparation | 3

31. Secondary Outcome: Number of Participants With On-Treatment Concomitant Nondrug Treatments/Procedures
Description: as for outcome 29
Time Frame: as for outcome 29
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants | 5

32. Secondary Outcome: Number of Participants With On-Treatment Concomitant Nondrug Treatments/Procedures by PT
Description: as for outcome 29
Time Frame: as for outcome 29
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Participants
  Abdominal cavity drainage | 2
  Bladder catheterisation | 1
  Endotracheal intubation | 1
  Enema administration | 1
  Enteral nutrition | 1
  Oxygen therapy | 1
  Platelet transfusion | 1
  Therapeutic procedure | 1
  Transfusion | 3

33. Secondary Outcome: Percentage of Participants Achieving Objective Response (OR) (Complete Response [CR] or Partial Response [PR]) (Confirmed or Unconfirmed)
Description: Tumor assessments were performed regularly during Cycles 1-12, then per local standard practice after Cycle 12. OR by investigator assessment was defined as a CR or PR according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 recorded from Cycle 1 Day 1 until disease progression, start of subsequent anti-cancer therapy or death due to any cause. CR is defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Short diameter is used in the sum for target nodes, while longest diameter is used in the sum for all other target lesions. An exact 95% confidence interval (CI) was calculated using Clopper-Pearson method. Given the exploratory nature of this endpoint, confirmation of response (CR/PR) was not required per protocol.
Time Frame: Cycle 1 Day 1 until disease progression, start of subsequent anti-cancer therapy or death due to any cause (maximum of approximately 45 weeks)
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 15
Percentage of participants | 6.7 [0.2 to 31.9]

34. Secondary Outcome: Duration of Response (DOR) for Participant(s) Achieving CR or PR
Description: Tumor assessments were performed regularly during Cycles 1-12 and per local standard practice after Cycle 12. Per RECIST v1.1, CR=complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions. Short diameter is used in the sum for target nodes, while longest diameter is used in the sum for all other target lesions. For participants with an OR (CR or PR), DOR = the time from first documentation of CR or PR to date of first documentation of objective progression or death. DOR data were censored on the date of last tumor assessment on study for participants who did not have objective tumor progression and who did not die due to any cause while on study. DOR was only calculated for participant(s) with an objective response. DOR was to be summarized using the Kaplan-Meier method if data permitted.
Time Frame: as for outcome 33
Population: The analysis population included all enrolled participants who received at least 1 dose of study intervention and had an objective response (CR or PR). Number of participants analyzed = number of participant(s) evaluable for this OM.
Measure: Number; unit: Days
Arm/Group | Talazoparib 1mg QD
Number analyzed (Participants) | 1
Days | 172

ADVERSE EVENTS:
Time Frame: From baseline (the latest non-missing value prior to or on the date of first dose of talazoparib) to at least 28 days after the last dose of talazoparib (maximum of 46 weeks)
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Talazoparib 1 mg QD
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=15)
Anaemia (Blood and lymphatic system disorders) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=15)
Anaemia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 4
Electrocardiogram T wave abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 6
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 3
White blood cell count decreased (Investigations) | 8
White blood cells urine positive (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT04635631/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04635631/SAP_001.pdf